CLINICAL TRIAL: NCT00845949
Title: Role of Chemokines and Proinflammatory Cytokines in Rheumatoid Synovial Pathological Changes
Status: Withdrawn | Type: Observational
Why Stopped: NO available budget and difficulty in recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chien-Sheng Wu, Chief, Division of Rheumatology, Far Eastern Memorial Hospital
Other Study IDs: 95034
Record Dates: First submitted 2008-03-03; First posted 2009-02-18 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Rheumatoid Arthritis
Keywords: chemokines synovium
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Synovial tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Rheumatoid arthritis is a common chronic destructive arthritis. Major pathology change in rheumatoid arthritis is synovium hyperplasia with bone and cartilage erosion. Infiltrates in synovial tissue included type one and type two synoviocytes, B cells, T cells and fibroblasts. These cells will release many cytokines and chemokines, which will induce expression of adhesion molecules, release of variable enzyme from fibroblast and osteoclast and result in bone erosion.

Recent study revealed that fibroblast-like synoviocytes (FLS) have some role in pathogenesis of rheumatoid arthritis.We believed CXCL12/CXCR4 ligand/receptor pair is important in chronicity of rheumatoid arthritis.

CXCL12 polymorphism is studied in many disease. There is no related CXCL12 polymorphism study in rheumatoid arthritis. Our study intended to clarify the relationship between pathology, serology factor, CXCL12 polymorphism in rheumatoid arthritis in hope that new direction of therapy will be elucidated.

DETAILED DESCRIPTION:
Rheumatoid arthritis is a common chronic destructive arthritis. Many patients suffered from disability from this disease. There is no satisfactory therapy for every patient. Present prognostic factor only explained the disease course partially.

Major pathology change in rheumatoid arthritis is synovium hyperplasia with bone and cartilage erosion. Infiltrates in synovial tissue included type one and type two synoviocytes, B cells, T cells and fibroblasts. These cells will release many cytokines and chemokines, which will induce expression of adhesion molecules, release of variable enzyme from fibroblast and osteoclast and result in bone erosion.

Previous study in rheumatoid arthritis focused mainly in role of lymphocytes and osteoclast. Recent study revealed that fibroblast-like synoviocytes (FLS) have some property which is similar but not identical to dendritic cells in lymph nodes. They are also important provider of IL-7 and IL-15 and play an important role in persisted activation of synovial tissue. Fibroblast will guide B cell infiltration and has intimate mutual interaction with T cells.

Stromal derived growth factor/CXCL12 is an effective lymphocyte chemokine. CXCR4 is corresponding receptor. CXCL12 has been associated with autoantibody production in lupus murine model animal. FLS can express stromal cell-derived factor 1 SDF-1/CXCL12, inducing persisted infiltration of CD4+ and CD8+ T cell. Furthermore, migration, proliferation and matrix mental proteinase secretion of FLSis regulated by CC and CXC chemokine. CXCL12 production by SLF is regulated by TNF-alpha, IL-1beta, and TGF-beta1, but there is still some inconsistency in literatures. CXCL12 itself also induce expression of CXCR4 and secretion of IL-6, IL-8 in FLS. Express of CCR4 in T cell is regulated by IL-2,IL-4,IL-7,IL-10 and cell contact. CXCL12 produced by SLF is also presented by endothelium cell and inducing angiogenesis. Clinical study also indicated that CXCL12 level is related to cartilage destruction. CXCL12 level is decreased after synovectomy. Therefore we believed CXCL12/CXCR4 ligand/receptor pair is important in chronicity of rheumatoid arthritis.

Recently CXCL12 polymorphism is studied in many disease, such as prognosis of HIV patients、chronic myeloproliferative disease, and AML metastasis. There is no related CXCL12 polymorphism study in rheumatoid arthritis. Our study intended to clarify the relationship between pathology, serology factor, CXCL12 polymorphism in rheumatoid arthritis in hope that new direction of therapy will be elucidated.

ELIGIBILITY:
Inclusion Criteria:

* patients with rheumatoid arthritis fulfills ACR 1987 classification criteria for rheumatoid arthritis

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Synovial tissue from patient with rheumatoid arthritis who underwent total knee replacement surgery after informed consent.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-11; Primary Completion 2008-06 (Estimated); Study Completion 2008-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Sheng Wu, Principal Investigator — Division of Allergy, Autimmunity and Rheumatology, Department of Internal Medicine
Locations (1):
- Division of Allergy, Autoimmunity and Rheuamtology, Department of Internal Medicine, Far Eastern Memorial Hospital, Banqiao District, Taiwan